CLINICAL TRIAL: NCT06119854
Title: Brief Digital Intervention to Increase COVID-19 Vaccination Among Individuals With Anxiety or Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City University of New York, School of Public Health (Other)
Collaborators: University of North Carolina, Chapel Hill (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Denis Nash, Professor, City University of New York, School of Public Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: RF1MH132360 (NIH); RF1MH132360 (NIH)
Record Dates: First submitted 2023-11-03; First posted 2023-11-07 (Actual); Results first posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Misinformation; Vaccine Hesitancy; Anxiety; Depression; COVID-19
Keywords: Anxiety; Depression; Vaccination; COVID-19
MeSH Terms: conditions — Communication; Vaccination Hesitancy; Anxiety Disorders; Depression; COVID-19

STUDY DESIGN:
Intervention Model Description: The investigators will assign undervaccinated cohort participants, with and without symptoms of anxiety or depression, to: 1) an attitudinal inoculation intervention; 2), a CBT-informed intervention; or 3) a conventional public health messaging intervention. Participants will be randomly assigned to one of the three intervention arms at a ratio of 1:1:1. Each arm will also be stratified 1:1 by presence or absence of anxiety or depression symptoms. Masking of participants to study arm assignment is not feasible due to the nature of the interventions. However, data collection analysts, study staff, and investigators will be masked to study arm assignments until analyses are complete.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Attitudinal inoculation intervention (Experimental): Participants randomized to this arm will view a brief video addressing one anti-vaccine "meta-narrative" or issue (e.g., concerns about the vaccine not working) most salient to the entire CHASING COVID study population (per recent historical data) and focused on bolstering resistance to mis/disinformation.
  Interventions: Behavioral: Attitudinal inoculation
- Cognitive behavioral therapy-informed intervention (Experimental): Participants randomized to this arm will view a brief video using a CBT-informed approach and focused on addressing barriers to vaccination, with no inoculation messaging.
  Interventions: Behavioral: Cognitive-behavioral therapy-informed intervention
- Conventional public health messaging (Active Comparator): Participants randomized to this arm will view a brief video conveying conventional public health messaging adapted from a review of public health public service announcements, with no inoculation or CBT-informed messaging.
  Interventions: Behavioral: Conventional public health messaging

INTERVENTIONS:
Behavioral: Attitudinal inoculation — A brief video focused on bolstering resistance to mis/disinformation about the COVID vaccine. Participants will receive two messages via text or email (1 and 3 days after the inoculation intervention). These messages will include reminders to get vaccinated.
  Arms: Attitudinal inoculation intervention
Behavioral: Cognitive-behavioral therapy-informed intervention — A brief video using a CBT-informed approach and focused on addressing barriers to COVID-19 vaccination. Participants will receive two messages via text or email (1 and 3 days after the inoculation intervention). These messages will include reminders to get vaccinated.
  Arms: Cognitive behavioral therapy-informed intervention
Behavioral: Conventional public health messaging — A brief video conveying conventional public health messaging adapted from a review of public health public service announcements with no inoculation messaging. Participants will receive two messages via text or email (1 and 3 days after the inoculation intervention). These messages will include reminders to get vaccinated.
  Arms: Conventional public health messaging

SUMMARY:
The COVID-19 pandemic has led to a mis/disinformation ecosystem that promotes divergent views of vaccine efficacy, as well as the legitimacy of science and medicine. Individuals are confronted with vaccine-related information from a multitude of sources, posing a challenge to identifying inaccurate information. COVID-19 vaccine uptake is lower among people with anxiety and depression than in the general population, due in part to higher levels of vaccine hesitancy. The prevalence of anxiety and depressive symptoms among US adults increased significantly during the COVID pandemic and has remained elevated. Interventions capable of mitigating the impact of vaccine hesitancy and mis/disinformation among undervaccinated people with anxiety or depression are therefore an urgent priority. Emerging evidence suggests that reasons for vaccine hesitancy and the impact of conventional vaccination messaging differ between those with and without mental health symptoms. There may also be added challenges overcoming logistical barriers to vaccination for people with anxiety or depressive symptoms.

The investigators aim to determine the effectiveness of two different brief digital intervention strategies compared with conventional public health messaging for increasing vaccine uptake in undervaccinated adults with and without anxiety or depressive symptoms. Attitudinal inoculation is a brief, scalable strategy that leverages the power of narrative, values, and emotion to strengthen resistance to mis/disinformation and reduce hesitancy. Though this approach has been shown to decrease COVID-19 vaccine hesitancy among US adults, the extent to which this approach increases COVID-19 vaccination remains unknown. Cognitive-behavioral therapy (CBT) is an evidence-based intervention for anxiety and depression. However, the efficacy of incorporating CBT-informed messaging in a vaccine promotion intervention has not been tested. The investigators hypothesize that both attitudinal inoculation and CBT-style communication will be more effective than conventional public health messaging to increase COVID-19 vaccination. The investigators also hypothesize that the CBT-informed intervention will be more effective than the attitudinal inoculation intervention for increasing COVID-19 vaccination among participants with symptoms of anxiety or depression.

DETAILED DESCRIPTION:
The project will recruit undervaccinated participants with and without symptoms of anxiety or depression from the CHASING COVID Cohort, a large and geographically diverse community-based US cohort, to tailor and test the effectiveness of two brief digital interventions to increase vaccine uptake among adults with anxiety or depressive symptoms. The investigators will assign undervaccinated cohort participants, with and without symptoms of anxiety or depression, to: 1) an attitudinal inoculation intervention; 2), a CBT-informed intervention; or 3) a conventional public health messaging intervention without attitudinal inoculation or CBT-informed content. The investigators will examine the outcome of COVID-19 vaccination at 4 weeks post-intervention, conducting intent-to-treat comparisons between arms.

ELIGIBILITY:
Inclusion Criteria:

* Recently engaged in the CHASING COVID Cohort study (i.e., started ≥ 1 survey since December 7, 2022)
* Last COVID-19 vaccine dose prior to September 11, 2023
* Current residence in the US or a US territory
* Comprehension of written English

Exclusion Criteria:

* No dose of a COVID-19 vaccine
* Had a SARS-CoV-2 infection in the past 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1419 (Actual)
Dates: Start 2024-04-15 (Actual); Primary Completion 2024-06-13 (Actual); Study Completion 2024-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Denis Nash, PhD, Principal Investigator — CUNY Institute for Implementation Science in Population Health
Locations (1):
- CUNY Graduate School of Public Health & Health Policy, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
CUNY Institute for Implementation Science in Population Health staff are available to assist externa researchers who may have further specific data questions or uses.

REFERENCES:
- [Background] Piltch-Loeb R, Su M, Hughes B, Testa M, Goldberg B, Braddock K, Miller-Idriss C, Maturo V, Savoia E. Testing the Efficacy of Attitudinal Inoculation Videos to Enhance COVID-19 Vaccine Acceptance: Quasi-Experimental Intervention Trial. JMIR Public Health Surveill. 2022 Jun 20;8(6):e34615. doi: 10.2196/34615. PMID 35483050
- [Background] Robertson MM, Kulkarni SG, Rane M, Kochhar S, Berry A, Chang M, Mirzayi C, You W, Maroko A, Zimba R, Westmoreland D, Grov C, Parcesepe AM, Waldron L, Nash D; CHASING COVID Cohort Study Team. Cohort profile: a national, community-based prospective cohort study of SARS-CoV-2 pandemic outcomes in the USA-the CHASING COVID Cohort study. BMJ Open. 2021 Sep 21;11(9):e048778. doi: 10.1136/bmjopen-2021-048778. PMID 34548354
- [Background] Parcesepe AM, Robertson M, Berry A, Maroko A, Zimba R, Grov C, Westmoreland D, Kulkarni S, Rane M, Salgado-You W, Mirzayi C, Waldron L, Nash D. The relationship between anxiety, health, and potential stressors among adults in the United States during the COVID-19 pandemic. medRxiv [Preprint]. 2020 Nov 4:2020.10.30.20221440. doi: 10.1101/2020.10.30.20221440. PMID 33173880
- [Derived] Piltch-Loeb R, Shen Y, Fleary S, Robertson M, Nunez Sahr J, Penrose K, Sanborn J, Yadav S, Srivastava A, Nash D, Parcesepe A. Testing Theory-Enhanced Messaging to Promote COVID-19 Vaccination Among Adults: Randomized Controlled Trial. J Med Internet Res. 2025 Oct 7;27:e79228. doi: 10.2196/79228. PMID 41057045

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Overall, 2,411 CHASING COVID Cohort participants were invited, and 1,419 (59%) were eligible and randomized to the intervention. After completing the 4-week survey, 16 participants were removed from the sample based on data quality protocols, leaving an analytic sample of 1403 participants. Randomization resulted in 469 individuals in CBT-kernels arm, 466 in the Inoculation arm, and 468 in the Standard public health messaging arm
Period: Overall Study
Arm/Group | Attitudinal Inoculation Intervention | Cognitive Behavioral Therapy-informed Intervention | Conventional Public Health Messaging
Started | 472 | 473 | 474
Completed | 466 | 469 | 468
Not Completed | 6 | 4 | 6

BASELINE CHARACTERISTICS:
Population: Overall, 2,411 CHASING COVID Cohort participants were invited, and 1,419 (59%) were eligible and randomized to the intervention. After completing the 4-week survey, 16 participants were removed from the sample based on data quality protocols, leaving an analytic sample of 1403 participants.
  Randomization resulted in 469 individuals in CBT-kernels arm, 466 in the Inoculation arm, and 468 in the Standard public health messaging arm (Figure 1).
Groups:
- Total: Total of all reporting groups
Arm/Group | Attitudinal Inoculation Intervention | Cognitive Behavioral Therapy-informed Intervention | Conventional Public Health Messaging | Total
Number analyzed (Participants) | 466 | 469 | 468 | 1403
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 415 | 416 | 415 | 1246
  >=65 years | 51 | 53 | 53 | 157
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender : Male | 183 | 192 | 199 | 574
  Gender : Female | 263 | 270 | 254 | 787
  Gender : Non-binary | 20 | 7 | 15 | 42
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Hispanic | 78 | 84 | 84 | 246
  Race/Ethnicity: White (non-Hispanic) | 268 | 288 | 286 | 842
  Race/Ethnicity: Black (non-Hispanic) | 60 | 49 | 42 | 151
  Race/Ethnicity: Asian/American Indian/Pacific (non-Hispanic) | 46 | 34 | 40 | 120
  Race/Ethnicity: Other/unknown | 14 | 14 | 16 | 44
Region of Enrollment [Count of Participants; unit: Participants]
  United States: MidWest | 72 | 76 | 84 | 232
  United States: NorthEast | 113 | 127 | 134 | 374
  United States: South | 167 | 163 | 135 | 465
  United States: Other | 1 | 1 | 1 | 3
  United States: West | 113 | 102 | 114 | 329
Number of COVID-19 vaccine doses as of Dec 2023 [Median (Inter-Quartile Range); unit: vaccine doses] — The total number of SARS-CoV-2 vaccination doses participants reported receiving as of the last CHASING COVID cohort assessment in December 2023
  vaccine doses | 3.00 [2.00 to 4.00] | 3.00 [2.00 to 4.00] | 3.00 [2.00 to 4.00] | 3.00 [2.00 to 4.00]

OUTCOME MEASURES:

1. Primary Outcome: Self-reported Receipt of COVID Vaccine Dose by 4 Weeks Post-intervention
Description: Following our theoretical premise that our intervention will impact the uptake of COVID-19 vaccination, the investigators define our primary outcome as self-reported receipt of a COVID vaccine dose in the 4 weeks post-intervention. Risk ratios will be used to estimate and compare the proportion of participants in each arm who achieved the outcome. The investigators will adjust for differences in measured pre-baseline variables to address potential imbalances and conduct a mediation analysis to better understand the intervention's mechanisms of action.
Time Frame: 4 weeks post-intervention
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Attitudinal Inoculation Intervention | Cognitive Behavioral Therapy-informed Intervention | Conventional Public Health Messaging
Number analyzed (Participants) | 466 | 469 | 468
Participants
  Received vaccine | 4 | 7 | 6
  Did not receive vaccine | 462 | 462 | 462
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy-informed Intervention vs Conventional Public Health Messaging; Test type: Other; Risk Ratio (RR) = 1.207, 95% CI 2-sided [0.406 to 3.590] — The CBT arm is the numerator and the standard arm is the denominator
Statistical Analysis 2: Comparison: Cognitive Behavioral Therapy-informed Intervention vs Conventional Public Health Messaging; Test type: Other; Risk Difference (RD) = 0.003, 95% CI 2-sided [-0.013 to 0.018] — RD was calculated as the risk in the CBT arm minus the risk in the standard arm
Statistical Analysis 3: Comparison: Attitudinal Inoculation Intervention vs Conventional Public Health Messaging; Test type: Other; Risk Ratio (RR) = 0.687, 95% CI 2-sided [0.194 to 2.436] — The inoculation arm is the numerator and the standard arm is the denominator
Statistical Analysis 4: Comparison: Attitudinal Inoculation Intervention vs Conventional Public Health Messaging; Test type: Other; Risk Difference (RD) = -0.004, 95% CI 2-sided [-0.018 to 0.010] — RD was calculated as the risk in the inoculation arm minus the risk in the standard arm

2. Secondary Outcome: Participants Classified as Vaccine Willing
Description: The investigators will estimate vaccine hesitancy at baseline, immediately post-intervention, 4 weeks post-intervention, and at 6 months post-intervention. People who indicate that they are "not willing" to get a vaccine dose will be defined as vaccine resistant, people who indicate that they are "somewhat willing" will be described as vaccine hesitant, and people who report that they are "very willing" or who report having received a vaccine dose will be classified as vaccine willing. Risk ratios will be used to estimate and compare the proportion of participants in each arm who are either vaccine resistant or vaccine hesitant to those who are vaccine willing at each time point. The investigators will adjust for differences in measured pre-baseline variables to address potential imbalances.
Time Frame: 4 weeks post-intervention
Population: Of the 1,403 participants analyzed at baseline, 59 participants were lost to follow up (20 in CBT arm, 21 in inoculation arm, and 18 in standard arm)
Measure: Count of Participants; unit: Participants
Arm/Group | Attitudinal Inoculation Intervention | Cognitive Behavioral Therapy-informed Intervention | Conventional Public Health Messaging
Number analyzed (Participants) | 445 | 449 | 450
Participants | 168 | 138 | 139
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy-informed Intervention vs Conventional Public Health Messaging; Test type: Other; Risk Ratio (RR) = 0.992, 95% CI 2-sided [0.785 to 1.253] — The CBT arm is the numerator and the standard arm is the denominator
Statistical Analysis 2: Comparison: Cognitive Behavioral Therapy-informed Intervention vs Conventional Public Health Messaging; Test type: Other; Risk Difference (RD) = -0.003, 95% CI 2-sided [-0.063 to 0.058] — RD was calculated as the risk in the CBT arm minus the risk in the standard arm
Statistical Analysis 3: Comparison: Attitudinal Inoculation Intervention vs Conventional Public Health Messaging; Test type: Other; Risk Ratio (RR) = 1.227, 95% CI 2-sided [0.981 to 1.534] — The inoculation arm is the numerator and the standard arm is the denominator
Statistical Analysis 4: Comparison: Attitudinal Inoculation Intervention vs Conventional Public Health Messaging; Test type: Other; Risk Difference (RD) = 0.070, 95% CI 2-sided [0.008 to 0.133] — RD was calculated as the risk in the inoculation arm minus the risk in the standard arm

3. Secondary Outcome: Self-reported Receipt of a COVID Vaccine Dose by 6 Months Post-intervention
Description: The investigators define our outcome as self-reported receipt of a COVID vaccine dose in the 6 months post-intervention. Risk ratios will be used to estimate and compare the proportion of participants in each arm who achieved the outcome. The investigators will adjust for differences in measured pre-baseline variables to address potential imbalances and conduct a mediation analysis to attempt to better understand the intervention's mechanisms of action.
Time Frame: 6 months post-intervention
Population: Of the 1,403 participants analyzed, 74 were lost to follow up by month 6 (25 in CBT arm, 23 in inoculation arm, and 26 in standard arm)
Measure: Count of Participants; unit: Participants
Arm/Group | Attitudinal Inoculation Intervention | Cognitive Behavioral Therapy-informed Intervention | Conventional Public Health Messaging
Number analyzed (Participants) | 443 | 444 | 411
Participants | 72 | 61 | 57
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy-informed Intervention vs Conventional Public Health Messaging; Test type: Other; Risk Ratio (RR) = 1.063, 95% CI 2-sided [0.740 to 1.527] — CBT group represents the numerator and standard (conventional) represents the denominator
Statistical Analysis 2: Comparison: Cognitive Behavioral Therapy-informed Intervention vs Conventional Public Health Messaging; Test type: Other; Risk Difference (RD) = 0.008, 95% CI 2-sided [-0.037 to 0.053] — RD was calculated as the risk in the CBT arm minus the risk in the standard arm
Statistical Analysis 3: Comparison: Attitudinal Inoculation Intervention vs Conventional Public Health Messaging; Test type: Other; Risk Ratio (RR) = 1.262, 95% CI 2-sided [0.892 to 1.784] — The inoculation arm is the numerator and the standard arm is the denominator
Statistical Analysis 4: Comparison: Attitudinal Inoculation Intervention vs Conventional Public Health Messaging; Test type: Other; Risk Difference (RD) = 0.034, 95% CI 2-sided [-0.013 to 0.080] — RD was calculated as the risk in the inoculation arm minus the risk in the standard arm

4. Secondary Outcome: Vaccine Willingness Post-intervention
Description: as for outcome 2
Time Frame: 6-months post-intervention
Population: Of the 1,403 participants analyzed at baseline, 76 participants were lost to follow up by month 6 (26 in CBT arm, 23 in inoculation arm, and 27 in standard arm)
Measure: Count of Participants; unit: Participants
Arm/Group | Attitudinal Inoculation Intervention | Cognitive Behavioral Therapy-informed Intervention | Conventional Public Health Messaging
Number analyzed (Participants) | 443 | 443 | 441
Participants | 202 | 172 | 152
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy-informed Intervention vs Conventional Public Health Messaging; Test type: Other; Risk Ratio (RR) = 1.131, 95% CI 2-sided [0.911 to 1.406] — CBT arm is the numerator and the standard arm is the denominator
Statistical Analysis 2: Comparison: Cognitive Behavioral Therapy-informed Intervention vs Conventional Public Health Messaging; Test type: Other; Risk Difference (RD) = 0.045, 95% CI 2-sided [-0.019 to 0.109] — RD was calculated as the risk in the CBT arm minus the risk in the standard arm
Statistical Analysis 3: Comparison: Attitudinal Inoculation Intervention vs Conventional Public Health Messaging; Test type: Other; Risk Ratio (RR) = 1.323, 95% CI 2-sided [1.074 to 1.631] — the inoculation arm is the numerator and the standard arm is the denominator
Statistical Analysis 4: Comparison: Attitudinal Inoculation Intervention vs Conventional Public Health Messaging; Test type: Other; Risk Difference (RD) = 0.111, 95% CI 2-sided [0.045 to 0.176] — RD was calculated as the risk in the inoculation arm minus the risk in the standard arm

5. Secondary Outcome: Vaccine Willingness Post-intervention
Description: as for outcome 2
Time Frame: immediately post-intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Attitudinal Inoculation Intervention | Cognitive Behavioral Therapy-informed Intervention | Conventional Public Health Messaging
Number analyzed (Participants) | 466 | 469 | 468
Participants | 153 | 133 | 141

ADVERSE EVENTS:
Time Frame: Adverse events were collected for 6 months after the intervention.
Arm/Group | Attitudinal Inoculation Intervention | Cognitive Behavioral Therapy-informed Intervention | Conventional Public Health Messaging
All-Cause Mortality (participants affected / at risk) | 0/466 | 0/469 | 0/468
Serious Adverse Events (participants affected / at risk) | 0/466 | 0/469 | 0/468
Other Adverse Events (participants affected / at risk) | 0/466 | 0/469 | 0/468

LIMITATIONS AND CAVEATS:
The study was conducted during a period of low COVID-19 activity, which may have reduced vaccine uptake. The brief video interventions may have limited impact, and participants were not required to watch them in full. Conducted late in the pandemic, findings may not generalize to earlier periods or future contexts. Follow-up is planned to assess longer-term effects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-05-02): https://cdn.clinicaltrials.gov/large-docs/54/NCT06119854/Prot_SAP_000.pdf